CLINICAL TRIAL: NCT00997464
Title: An Exploration of Factors Affecting Interest and Uptake of Genetic Testing for Prostate Cancer Susceptibility: The Clinical Application of Genetic Testing for Lower Risk Cancer Predisposition Genes
Brief Title: An Exploration of Genetic Testing for Prostate Cancer Susceptibility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Dr. Rosalind Eeles, Institute of Cancer Research
Other Study IDs: CCR3200
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study of the factors that affect interest in - and uptake of - genetic testing for variants that predispose to prostate cancer from the perspective of the patient.

DETAILED DESCRIPTION:
This study will use a mixed methods approach to follow men as they move through the genetic testing process, from initial contact through to receiving their genetic testing results. A questionnaire will be used to measure variables at both baseline and after proceeding through the testing process. A small cohort of men will be invited to be interviewed to gather some in depth qualitative data about the issues that have arisen during the study process.

ELIGIBILITY:
Inclusion Criteria:

* Men with a positive family history of prostate cancer. The definition of a positive family history will be: Men with a first degree relative with prostate cancer diagnosed at <70 years; Men with two relatives with prostate cancer where at least on is diagnosed at <70 years; Men with three relatives with prostate cancer diagnosed at any age
* Age 40-69 years
* No previous biopsy for raised PSA
* Absence of any psychological, familial, sociological or geographic situation potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

* Previous prostate cancer
* Men from families where there is known to be a mutation in a high-risk prostate cancer gene
* Men who have had a prostate biopsy within the last 12 months.

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men with strong family history of prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Whether cancer worry changes between the two time-points (measured using the Impact of Event Scale)

SECONDARY OUTCOMES:
Why are men interested/ not interested in seeking genetic profiling for prostate cancer, and what might be the uptake of such testing?
What are the expectations of this testing from the perspective of the user, what are the perceived benefits and limitations of testing and how do these change through the testing process
Is there a relationship between a family history of cancer, cancer worry, and a persons intention to seek genetic testing?
How would the information provided by such a test be used by the individual and the family and how could this impact upon the healthcare system

CONTACTS AND LOCATIONS:
Overall Officials: Dr Rosalind Eeles, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom